CLINICAL TRIAL: NCT00987701
Title: Correlation Between Perineuraxial Anesthesia Fluid Resuscitation in Cesarean Section and Infant Neurobehaviors
Brief Title: Perineuraxial Anesthesia Fluid Management and Infant Neurobehaviors
Acronym: PAFUMIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NJMU-0932MZ; NMUK2190
Record Dates: First submitted 2009-09-30; First posted 2009-10-01 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Cesarean Section
Keywords: Neurobehavior; Development; Fluid management; Neuraxial anesthesia
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Crystalloid resuscitation (Active Comparator): Crystalloid (Ringer's lactate) will be delivered before (15min) or after (15min) neuraxial anesthesia
  Interventions: Drug: Ringer's Lactate
- Colloid resuscitation (Active Comparator): Colloid (6% hydroxyethyl starch ) will be delivered before (15min) or after (15min) neuraxial anesthesia
  Interventions: Drug: Six percent hydroxyethyl starch

INTERVENTIONS:
Drug: Ringer's Lactate — Ringer's Lactate 8 ml/kg was given intravenously before or after epidural, spinal or CSEA in cesarean section
  Other Names: Lactated Ringer's solution
  Arms: Crystalloid resuscitation
Drug: Six percent hydroxyethyl starch — Hydroxyethyl starch (6%) was given before or after epidural, spinal or CSEA in cesarean section
  Other Names: HES/HAES
  Arms: Colloid resuscitation

SUMMARY:
Early change in neurobehavior is strongly associated with the intelligence development of children. Previous studies reported that cesarean section itself could influence the later development of children. In addition, neuraxial anesthesia including epidural, spinal and combined spinal epidural anesthesia (CSEA) are the major forms used during cesarean delivery, and these anesthesia techniques will undoubtedly evoke hypotension and corresponding hemodynamic alteration, of which would result in decreasing in umbilical placental insufficiency and fetus hypoxia leading to early abnormality of neurobehaviors in infants. Fluid management, such as crystalloid and colloid, is the common ones given before or / and after neuraxial anesthesia to prevent or reverse hypotension. However, it is still unknown whether the perineuraxial anesthesia fluid resuscitation could improve the neurobehavior scorings, and could produce positive effect on later intelligence development. Herein the investigators hypothesized that effective perineuraxial anesthesia fluid management during cesarean section would prevent the occurrence of hypotension and improve infant's neurobehavior scorings.

ELIGIBILITY:
Inclusion Criteria:

* 21-40 yr
* First time of delivery
* ASA status I-II
* No premature
* No genetic and infectious diseases
* Chinese

Exclusion Criteria:

* < 21 yr
* > 40 yr
* Subjects with cardiac and pulmonary disorders
* Dislocation of placenta
* Pregnant hypertension
* Allergy to local anesthetics
* Unwilling to cooperation
* With significant delivery side effects

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5000 (Actual)
Dates: Start 2009-09; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | Immediate after birth (0 min)

SECONDARY OUTCOMES:
Apgar scoring | One min and 5min after birth.
Umbilical-cord gases analysis | At the time baby was born (0min)
Neonatal sepsis evaluation | One hour after the baby was born
Neonatal antibiotic treatment | One hour after the baby was born
Incidence of maternal side effects | Analgesia initiation (0min) to successful vaginal delivery (this time encountered alteration with different women)
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 30min after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1h after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 8h after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1d after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1wk after birth
Neurobehavior evaluation with the Assessment of Preterm Infants' Behavior (APIB) | 1month after birth

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- The Affiliated Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu, China